CLINICAL TRIAL: NCT06642922
Title: Correlation Between BMI , Balance and Gross Motor Capacities in Children with Spastic Diplegia
Brief Title: Gross Motor Abnormalities in Relation to Balance and Weight Indicators in Diplegia
Acronym: BMI
Status: Completed | Type: Observational
Sponsor: Lamis Neyazy Elrakhawy (Other)
Responsible Party: Sponsor-Investigator, Lamis Neyazy Elrakhawy, principal investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.REC/012/004585; faculty of physical therapy (Registry Identifier: P.T.REC/012/004585)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2021-08

CONDITIONS: Spastic Diplegia Cerebral Palsy
Keywords: BMI; Balance; Gross motor capacities; obesity; diplegia
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group 1: normal weight group , 53 participants BMI , balance , and gross motor capacities were assessed for each participant
- group 2: overweight and obese group , 51 participants BMI , balance , and gross motor capacities were assessed for each participant

SUMMARY:
The goal of this observational study is to investigate the correlation between BMI and balance and gross motor capacities in children with spastic diplegia. The main question it aims to answer is:

Is there a correlation between BMI, balance disturbances and gross motor capacity in children with spastic diplegic cerebral palsy? Researchers compared between results of biodex balance system , GMFM and BMI measures participants stood on biodex balance platform for balance measurement and performed Gross Motor Function Measurement items for gross motor capacities assessment

DETAILED DESCRIPTION:
Spastic diplegia is the most common type of CP that results in problems with posture, balance, as well as gait control. For children suffering from spastic diplegic CP, balance problems provide a significant difficulty since they make it difficult for them to achieve and maintain balance . Additionally, they commonly demonstrate delayed development of gross motor function that has been connected to functional outcomes, such as daily living tasks . The prevalence of obesity in the CP population has risen over the last decade from 7.7 to 16.5 %. . Obesity is associated with health risks and difficulties in balance and walking. this cross-sectional-correlation study was conducted at the Outpatient Clinic at the Faculty of Physical Therapy, Cairo University. The study included 104 diplegic children aged from 5-10 years, 53 in normal weight group and 51 in overweight group. Dynamic balance was evaluated by overall stability index (OSI) in biodex balance system and gross motor capacities (GMC) were evaluated by standing &walking dimensions in GMFM

ELIGIBILITY:
Inclusion Criteria:

Children selected according to the following criteria:

* Diagnosed with diplegic CP
* Their ages will range between 5 and 10 years
* Subjects will participate according to BMI classification ; normal weight in the first group and (obese , overweight) in the second group .
* They must be able to stand independently.
* Have minimum height of 100 cm.
* Have a developmental level of grade I or II according to gross motor function classification system GMFM.
* Able to understand and follow instructions.

Exclusion Criteria:

* Auditory defects.
* Visual defects.
* Cognitive or vestibular defects.
* Use of an assistive device.
* Fixed deformity, bony or joint limitation.
* Surgery (tendon lengthening).

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with spastic diplegia aged from 5 to 10 years old
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
BMI | 9 months
  Standardized height-weight measuring scale for measurement of weight and height, to be able to calculate BMI Growth charts were used to plot BMI and age separately for girls and boys. Then, each subject was given a percentile and put into one of two categories: normal (5th to 85th percentile) and overweight, obese (85th and above percentile).
balance assessment | 9 months
  Biodex balance system SD with movable platform was used .The overall stability index (OSI) will be measured as indicator of dynamic balance. The higher the OSI values, the lower the dynamic balance stability. Bilateral stance (standing on both legs), eyes open, stability level 5 (12 is the most stable level), and three repeated trials (for more accuracy) for 20 seconds (test time for each trial) were the test conditions

SECONDARY OUTCOMES:
gross motor capacities | 9 months
  GMC assessed by using dimensions D and E of the Gross Motor Function Measure (GMFM-88) which measures respectively activities in standing, and walking, running, and jumping. . A 4-point scale was used and scores were expressed as percentages

CONTACTS AND LOCATIONS:
Overall Officials: khaled A Mamdouh, Principal Investigator — Department of Physical Therapy for Pediatrics, Faculty of Physical Therapy, Cairo University; Hoda A Eltalawy, Study Director — Department of Physical Therapy for Pediatrics, Faculty of Physical Therapy, Cairo University; Radwa s Abdulrahman, Study Director — Department of Physical Therapy for Pediatrics, Faculty of Physical Therapy, Cairo University
Locations (1):
- Lamis Neyazy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No